CLINICAL TRIAL: NCT06740253
Title: Safety and Acceptability Study of MM008-IVR, an Antibody-Based Nonhormonal Contraceptive Intravaginal Ring
Brief Title: Safety and Acceptability Study of a Placebo Antibody-Based Nonhormonal Contraceptive Intravaginal Ring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: Mucommune, LLC. (Unknown); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 24-0194; 1R43HD108823-01 (NIH)
Record Dates: First submitted 2024-11-25; First posted 2024-12-18 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Healthy Female Subjects
Keywords: Non-hormonal intravaginal ring

STUDY DESIGN:
Intervention Model Description: Study participants will be asked to use a placebo IVR to determine safety and acceptability for 14 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Placebo IVR (Experimental): Participants will use a placebo IVR for 14 days.
  Interventions: Device: Placebo intravaginal ring (IVR)

INTERVENTIONS:
Device: Placebo intravaginal ring (IVR) — Antibody-Based Nonhormonal Placebo Contraceptive Intravaginal Ring

SUMMARY:
In order to deliver nonhormonal vaginal contraceptive using anti-sperm antibodies, a new vaginal ring design using a capsule-IVR will be utilized. Evaluating the safety and acceptability of this device early in the product development cycle is important, not only because device/formulation characteristics become increasingly difficult to alter as product is advanced into clinical trials, but also because user adherence can directly impact clinical trial outcomes.

DETAILED DESCRIPTION:
There is a gap in commercially available reliable, effective contraception methods that do not contain hormones. Mucommune is developing a novel non-hormonal contraceptive in the form of a capsule-intravaginal ring (IVR) that releases highly potent contraceptive antibodies (MM008) that rapidly bind and trap sperm. These antibodies have been developed over the past 5 years and the target on sperm cells was initially obtained from a patient with infertility due to anti-sperm antibodies.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent
2. Age of 18 - 45 years at enrollment
3. Female participants, born female
4. Willing and able to

   * communicate in English
   * complete all required study procedures
5. Subjects willing to abstain from vaginal intercourse and use of vaginal products for the first week of the study and until cleared by the study physician.

Exclusion Criteria:

Participant reports any of the following:

1. Gynecologic or genital procedure (e.g., tubal ligation, dilation and curettage, piercing) within 21 days prior to Enrollment Note: Colposcopy and cervical biopsies for evaluation of an abnormal Pap smear as well as IUD removal are not exclusionary
2. Current use of an IVR (e.g., Nuvaring)
3. Prior hysterectomy
4. Females who are pregnant based on positive pregnancy test by urine HCG
5. Cervicovaginal inflammation or epithelial disruption on colposcopy at the screening examination.
6. Current active gynecological abnormalities or sexually transmitted infection and/or vaginal pathogens (e.g. gonorrhea, chlamydia, mycoplasma genitalium, trichomonas, candida species, bacterial vaginosis) at the screening examination.

   Note: Subjects may be treated and re-screened for participation.
7. Has any other condition or is participating in another research study that, in the opinion of the Principal Investigator or designee, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving study objectives.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only female born subjects are eligible to participate.
Enrollment: 14 (Actual)
Dates: Start 2025-02-11 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2025-07-28 (Actual)

PRIMARY OUTCOMES:
Device Safety | 14 days
  Determined by AE's, including colposcopy findings, that are deemed to be product related during placebo IVR use.

SECONDARY OUTCOMES:
Device-only tolerability and acceptability | 14 days
  Device tolerability and acceptability as judged by scores on the questionnaires related to placebo IVR use. The scale that is used is a 5 point likert scale that assesses the degree to which the participant agrees or disagrees with a statement regarding the use of the intravaginal ring. Items will be factor analyzed and items will be summed by subscale with a higher score indicating greater agreement or a lower score indicating less agreement with a variety of statements about the ring and their experience of using the ring.

OTHER OUTCOMES:
Changes in pro-inflammatory cytokines | 14 Days
  Measures of proinflammatory cytokines at baseline and after placebo IVR use will be done using the ProcartaPlex Human Cytokine/Chemokine/Growth Factor Convenience Panel 1, 45plex. It allows for detection and quantification of up to 45 protein targets. This will be utilized to measure proinflammatory cytokines in the vaginal secretions. Increases in the proinflammatory cytokines indicate an increase in inflammation.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided